CLINICAL TRIAL: NCT06531746
Title: Effect of Extracorporeal Shock Wave on Electrophysiological Changes and Pain in Patients With Lower Cross Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahmed Alshimy (Other)
Responsible Party: Sponsor-Investigator, Ahmed Alshimy, Lecturer of Physical Therapy for Neurology and its Surgery Faculty of Physical Therapy - Al Ryada University for Science and Technology, AlRyada University for Science & Technology
Organization: AlRyada University for Science & Technology (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/005231
Record Dates: First submitted 2024-07-29; First posted 2024-08-01 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Lower Cross Syndrome
Keywords: Extracorporeal Shock Wave; Electrophysiological changes; Pain; Lower Cross Syndrome
MeSH Terms: conditions — Pain | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (I) (Experimental): Will consist of 20 patients with lower cross syndrome and will receive extracorporeal shock wave in addition to conventional physical therapy program. For 12 sessions every other day, each session for 1 hour.
  Interventions: Other: Extracorporeal shock wave; Other: Conventional physical therapy program
- Control group (II) (Experimental): Will consist of 20 patients with lower cross syndrome and will receive sham extracorporeal shock wave in addition to conventional physical therapy program only same as group (I). For 12 sessions every other day, each session for 1 hour.
  Interventions: Other: Conventional physical therapy program; Device: Sham (No Treatment)

INTERVENTIONS:
Other: Extracorporeal shock wave — participants will receive 2000 ESWT impulses, with 1500 targeting the taut band and 500 surrounding the taut band, with an energy flux density of 0.10 mJ/mm and frequency of 8 Hz, by using an
  EME S.r.l. via Degli Abeti 88/161122 Pesaro [serial number:
  EM12681015], Italy, shock wave generator.
  Arms: Study group (I)
Other: Conventional physical therapy program — Stretching and strengthening of Iliopoas muscle and Stretching and strengthening of Lower back muscles
Device: Sham (No Treatment) — Sham extracorporeal shock wave will be introduced without real shock wave impulses.
  Arms: Control group (II)

SUMMARY:
Lower Cross Syndrome happens when there is muscular imbalance between weak and tight muscles. The tight muscles are generally the hip flexors and erector spinae, and weak muscles are the abdominals and gluteal muscles. Shortening occurs in the hip flexors while weakening occurs in the abdominals and gluteal muscles.

DETAILED DESCRIPTION:
Group I (Study): will consist of 20 patients with lower cross syndrome and will receive extracorporeal shock wave in addition to conventional physical therapy program. For 12 sessions every other day, each session for 1 hour.

Group II (Control): will consist of 20 patients with lower cross syndrome and will receive sham extracorporeal shock wave in addition to conventional physical therapy program only same as group (I). For 12 sessions every other day, each session for 1 hour.

ELIGIBILITY:
Inclusion Criteria:

1. Forty-four lower cross syndrome patients from both genders their ages ranged from 30-45 years old.
2. All patients in present study will be ambulant independently.
3. All patients will be medically stable.
4. The body mass index (BMI) will be ranged from 20:25 Kg/m2.

Exclusion Criteria:

1. Patients with musculoskeletal deformities and disorders.
2. Patients with psychiatric disorders or seizures.
3. Patients with visual and auditory impairment or tremors influencing balance.
4. Patients with other neuromuscular disorders.
5. Patients with BMI more than 25 kg/m2.
6. Patients with cognitive impairment.
7. Patients with lower limb or head and brain surgeries.

Ages: 30 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2025-02-02 (Actual); Primary Completion 2025-11-28 (Actual); Study Completion 2025-11-29 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | 4 weeks
  Assess pain intensity
Electromyograph | 4 weeks
  Assess activity of lower back muscles (Erector Spinae)

CONTACTS AND LOCATIONS:
Locations (1):
- Al Ryada University for Science and Technology, Sadat, Menoufia, Egypt

IPD SHARING:
Plan to Share IPD: No